CLINICAL TRIAL: NCT06628206
Title: Phase 1b Randomized, Double Blind, Placebo-controlled Study to Evaluate Safety, Tolerability and Pharmacokinetics of LPX-TI641 in Patients With Rheumatoid Arthritis and Psoriatic Arthritis
Brief Title: Safety and Pharmacokinetics of LPX-TI641 in Rheumatoid Arthritis and Psoriatic Arthritis
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: LAPIX Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LPX641-102
Record Dates: First submitted 2024-09-26; First posted 2024-10-04 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-04

CONDITIONS: Rheumatoid Arthritis (RA); Psoriatic Arthritis (PsA)
Keywords: Phase 1 study; pharmacokinetics; safety
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis, Psoriatic

STUDY DESIGN:
Intervention Model Description: There will be 2 cohorts, one for each indication. Each cohort will consist of ~ 16-to-60 participants (Total ~up to 120 participants in the study). The first cohort is for RA and in this cohort the first 5 participants will receive LPX-TI641 at 60 mg QD (4 mg/mL formulation) or placebo for 28 days (randomized in 3:2 treatment:placebo). Subsequently, 3 RA participants will receive LPX-TI641 at 60 mg QD (16 mg/mL formulation, (non-randomized). The next 8 RA participants (randomized in 3:1 treatment:placebo) will receive LPX-TI641 at 120 mg QD (4 participants 4 mg/ml formulation and 4 participants 16 mg/ml formulation). The remaining participants in the RA cohort (up to 44 participants) will receive the compounded capsule formulation with 150 mg LPX-TI641 or placebo (3:1 treatment:placebo). The psoriatic arthritis cohort will receive the compounded capsule formulation with 150 mg LPX-TI641 or placebo. Overall, participants in both cohorts will be randomized in a 3:1 ratio.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Sponsor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Rheumatoid arthritis (Experimental): LPX-TI641 or Placebo
  Interventions: Drug: LPX-TI641; Drug: Placebo
- Psoriatic Arthritis (Experimental): LPX-TI641 or Placebo
  Interventions: Drug: LPX-TI641; Drug: Placebo

INTERVENTIONS:
Drug: LPX-TI641 — Oral administration QD for 28 consecutive days
Drug: Placebo — Drug is LPX-TI641. Placebo an identical formulation without the LPX-TI641.

SUMMARY:
The goal of this clinical trial is to study the drug LPX-TI641 in patients with rheumatoid arthritis and psoriatic arthritis. We will compare the safety and tolerability of LPX-TI641 to placebo that contains no drug. We will also evaluate the plasma pharmacokinetics of LPX-TI641. LPX-TI641 (or placebo) will be administered orally for 28 days.

DETAILED DESCRIPTION:
This is a Phase 1b, multi-center, randomized, double-blind, parallel-group, placebo-controlled multiple dose study in participants with rheumatological conditions (rheumatoid arthritis, psoriatic arthritis).

There will be 2 cohorts, one for each indication. Each cohort will consist of ~ 16-60 participants (Total ~up to 120 participants).

The Primary objective of the study is to evaluate the safety and tolerability after multiple oral doses of LPX-TI641 in participants with RA and PsA.

And the secondary objective of the study is to evaluate the plasma pharmacokinetics after multiple oral doses of LPX-TI641 in participants with RA and PsA.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has signed an Informed Consent Form (ICF) prior to any study-specific procedures being performed
2. ≥ 18 years old, irrespective of their race and ethnicity.
3. Body Mass Index (BMI) 18.0-35.0 kg/m2, inclusive, at screening.
4. Participants are willing and able to adhere to study protocol requirements including but not limited to scheduled outpatient visits, inpatient hospital stay, laboratory tests, and 12-lead ECGs.
5. A. Diagnosis of RA and meeting the 2010 American College of Rheumatology (ACR)/European League Against Rheumatism (EULAR) classification criteria for RA at least 3 months prior to screening AND Active disease defined by ≥ 6 tender out of 68 joints and ≥ 6 swollen out of 66 swollen joint count at both screening and Day 1.

   AND Participants received conventional synthetic disease-modifying antirheumatic drug (csDMARD) therapy for ≥ 3 months and on a stable dose for ≥ 4 weeks prior to the first dose of study drug. The csDMARD allowed include methotrexate (MTX) (≤ 25mg/week), sulfasalazine (3 grams a day), hydroxychloroquine (≤400mg/day), chloroquine (≤250mg/day), and leflunomide (≤ 20mg/day) or intolerance to csDMARD as assessed by the investigator OR B. PsA diagnosis of at least 3 months duration prior to the date of first screening with Classification of Psoriatic Arthritis (CASPAR) confirmed diagnosis at Screening. Have active psoriasis defined by at least 1 psoriasis lesion >= 2 cm diameter in areas other than the axilla or groin.

   AND Active disease defined by ≥ 3 tender out of 68 joints and ≥ 3 swollen out of 66 swollen joint count at both screening and Day 1.

   AND Participants received standard doses of NSAIDS for ≥4 weeks or csDMARDS (MTX ≤ 25mg/week), sulfasalazine (3 grams a day), and leflunomide (≤ 20mg/day), administered for ≥ 3 months and on a stable dose for ≥ 4 weeks prior to the first dose of study drug or intolerance to NSAIDS or DMARDs as assessed by the investigator. Other traditional DMARDS not listed as a prohibited concomitant medication may be considered after discussion with the Study physician.
6. The subject must be judged to be in good health by the investigator to participate in the study, based on clinical evaluations, including laboratory safety tests, medical history, physical examination, vital signs and 12-lead ECG competed at the screening visit and prior to the first dose of study drug.
7. Female subject is postmenopausal (at least 1 year; to be confirmed by follicle stimulating hormone (FSH) if less than 2 years since last menstrual period), permanently sterilized (e.g. tubal occlusion, hysterectomy, bilateral salpingectomy or if of childbearing potential and engaged in sexual activity that can result in pregnancy must agree to use any two of the highly effective contraception methods listed below. Male participants with a partner of childbearing potential must also agree to use any two of the highly effective contraception methods listed below between the both of them. This criterion must be followed from screening visit to 6 weeks after the last dose in females and for 90 days after the last dose for males.

   a. The following applies to all female participants with childbearing potential and female partners of male volunteers enrolled in the study.

   i. Implantable progestogen-only hormone contraception associated with inhibition of ovulation.

   ii. Intrauterine device. iii. Intrauterine hormone-releasing system. iv. Bilateral tubal occlusion. v. Combined (estrogen- and progestogen-containing) hormonal contraception associated with inhibition of ovulation:
   1. Oral
   2. Intravaginal
   3. Transdermal
   4. Injectable vi. Progestogen-only hormone contraception (oral or injectable) is associated with inhibition of ovulation.

   vii. Vasectomized partner viii. Sexual abstinence -this is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study intervention. The reliability of sexual abstinence needs to be evaluated about the duration of the study and the preferred and usual lifestyle of the participant.

   ix. A combination of male condoms with either cervical cap, diaphragm, or sponge with spermicide (double-barrier methods) b. The following applies to all male participants in the study: i. Sexual abstinence- this is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study intervention. The reliability of sexual abstinence must be evaluated for the study and the participant's preferred and usual lifestyle.

   ii. A combination of male condoms with either cervical cap, diaphragm, or sponge with spermicide (double-barrier methods).

   iii. Vasectomy
8. Negative serum B-human chorionic gonadotropin test at screening (for all females) and negative urine pregnancy at randomization (Day 1) (females of childbearing potential) prior to administration of investigational product.

Exclusion Criteria:

* Any subject who meets any of the following criteria will not qualify for entry into the study:

  1. History of clinically significant medical conditions or any other reason that in the opinion of the PI would interfere with subject's participation in this study
  2. History of clinically significant per the PI's opinion drug or alcohol abuse within the last 6 months
  3. Pregnant or lactating women or women currently undergoing infertility treatments or women who intend to become pregnant during the time of study enrollment.
  4. Any known history of malignancy within 5 years other than other than completely treated non-metastatic basal cell carcinomas or squamous cell carcinomas of the skin or localized carcinoma in situ of the cervix.
  5. Any known history of a rheumatologic, autoimmune or cutaneous disease other than RA (except secondary Sjögren's syndrome), or PSA.
  6. Significant systemic involvement secondary to RA/PsA (active vasculitis, pulmonary fibrosis, or Felty's syndrome).
  7. Currently have non-plaque forms of psoriasis e.g. erythrodermic, guttate or pustular with the exception of nail psoriasis which is allowed.
  8. Receipt of an investigational therapy less than 3 months or 5 drug-elimination half-lives (whichever is longer) prior to first administration of study treatment and during the study
  9. Receipt of any of the following excluded therapies:

     Any cell depleting therapy including but limited to anti-CD4, anti-CD5, anti-CD3, rituximab, ocrelizumab, or ofatumumab.

     Have received prior tsDMARDs including but not limited to inhibitors of Janus kinase (JAK), Bruton tyrosine kinase, or tyrosine kinase 2, including baricitinib, tofacitinib, upadacitinib, filgotinib, ibrutinib, or fenebrutinib.

     Have received prior immunomodulatory bDMARDs including, but not limited to adalimumab, golimumab, ustekinumab, secukinumab, tocilizumab, abatacept, belimumab, anifrolumab or other inhibitors of TNF, IL-6, IL-23, or IL-17 Receipt of any other conventional DMARDs (not allowed per inclusion criteria 3) within less than 5 half-lives, prior to screening visit.
  10. Lack of response to > 1 therapeutic agent targeting tumor necrosis factor.
  11. If on prednisone, subject must be on stable dose, not to exceed equivalent of 10mg of prednisone per day (RA and PsA), and dose must be stable for ≥ 4 weeks prior to Day 1. No injected corticosteroids 8 weeks prior to first dose of study drug (e.g intraarticular, intramuscular, or intravenous)
  12. Use of psoriasis treatments:

      1. Oral or topical retinoids 2 weeks prior to Day 1 and throughout the study
      2. Topical treatments (steroids, or JAK inhibitors) within 2 weeks prior to Day 1 and throughout the study
      3. PUVA or UVB phototherapy within 4 weeks prior to Day 1 and throughout the study.
  13. No high potency opioid analgesics 2 weeks prior to baseline and during study. Analgesic dose must remain stable throughout from screening through completion of the study.
  14. COVID-19:

      The subject has COVID-19 positive status (confirmed by clinical signs and symptoms and a positive SARS-CoV-2 NAAT or rapid antigen COVID test) at any time during the screening period.

      OR has had recent COVID-19 vaccination including a booster dose in the past 30 days prior to screening OR has received anti-viral therapy intended to prevent COVID-19 such as nirmatrelvir/ritonavir, remdesivir, molnupiravir, interferons, anti-SARS-CoV-2 monoclonal antibodies, IVIG SARS-CoV-2, COVID-19 convalescent plasma, etc. within the past 30 days prior to screening
  15. Subject has clinical or laboratory evidence of active or latent tuberculosis (TB) infection at screening as assessed by QuantiFERON-TB-Gold or a purified protein derivative skin test or equivalent (or both if required per local guidelines) and chest X-ray. Chest X-rays taken within 2 months prior to screening may be used instead of during screening if there is documentation showing no evidence of infection or malignancy as read by qualified physician.
  16. Any active or recurrent infection within the past 4 weeks prior to screening requiring IV or oral antibiotics.
  17. Laboratory values of the following at the Screening Visit:

      Hemoglobin < 9 g/dL for males and < 8.5 g/dL for females WBC <3.5X109/L; Absolute neutrophil count (ANC) < 1500 cells/µL, (or < 1200 cells/µL for Black participants of African descent) Aspartate aminotransferase or alanine aminotransferase > 2.0 x the upper limit of normal (ULN) or bilirubin >= ULN; Bilirubin >ULN Serum creatinine > 1.5 x the ULN; Platelets < 100,000 cells/[mm^3] (10^9/L); Clinically significant abnormal screening laboratory results as evaluated by the Investigator
  18. Acutely worsened renal function within past 3 months prior to screening or estimated creatinine clearance <60ml/min by CKD-EPI creatinine equation
  19. Participants with a history of active or latent TB will be excluded from the study, unless documentation of complete TB treatment, consistent with local country guidelines, can be provided.
  20. Subject has any clinically significant finding on 12-lead ECG at screening or admission. NOTE: QTc(F) interval of >450 msec in male participants or >470 msec in female participants will be the basis for exclusion from the study. ECG may be repeated once for confirmatory purposes if initial values obtained exceed the limits specified.
  21. Subject with positive results for HBsAg (hepatitis B surface antigens) and/or HBcAb (Hepatitis B core antibodies) and/or HCV Ab (hepatitis C antibodies), and/or HIV Ab (human immunodeficiency virus antibodies).
  22. Blood loss of >250 mL or donated blood within 56 days or donated plasma within 7 days of screening.
  23. Recent vaccination with live attenuated vaccines such as influenza, measles, mumps, and rubella (MMR), Herpes zoster, varicella, yellow fever, Rotavirus vaccine, etc., or inactivated vaccines such as Hepatitis A, rabies vaccine, etc. in the past 30 days.
  24. History of infection 1) requiring hospitalization or parenteral antimicrobial therapy within 3 months prior to Day 1 or 2) treated with oral antimicrobial therapy within 2 weeks prior to Day 1.
  25. Subject is investigative site personnel, sponsor personnel, or a member of their immediate families (spouse, parent, child or sibling whether biological or legally adopted).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-12-15 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability after multiple oral doses of LPX-TI641 in participants with RA and PsA. | 56 days
  Rate and severity of treatment-emergent adverse events, including serious adverse events.

SECONDARY OUTCOMES:
To evaluate the plasma pharmacokinetics after multiple oral doses of LPX TI641 in participants with RA and PsA. | 24 hours on Day 1 and 24 hours on Day 28
  Measure Area Under the Concentration Time Curve after single dose and at Steady State
To evaluate the plasma pharmacokinetics after multiple oral doses of LPX TI641 in participants with RA and PsA | 24 hours on Day 1 and 24 hours on Day 28
  Measure maximum plasma concentration (Cmax) after single dose and at Steady State

CONTACTS AND LOCATIONS:
Locations (1):
- Triumpharma Clinical Research Unit at AlEssra Hospital, Amman, Jordan

IPD SHARING:
Plan to Share IPD: No